CLINICAL TRIAL: NCT01171755
Title: A Phase II Study of Gemcitabine and TS-1 in Patients With Previously Untreated Metastatic or Recurrent Biliary Tract Cancer
Brief Title: Phase II Study of Gemcitabine and TS-1 in Biliary Trat Cancer
Acronym: GetBil
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The objective response rate by more than two people are confirmed.
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-11-008; 82-02-3410-0914
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2012-01

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Ts-1 (Experimental): Gemcitabine : 1000/m2 will be administered on days 1 and 8 at every 3 weeks . TS-1 will be administered orally according to body surface area (BSA) as follows : BSA<1.25 M2, 80 mg/day; 1.25 M2≤BSA<1.5 M2, 100 mg/day; 1.5 M2≤BSA, 120 mg/day for 14 consecutive days followed by a 7-day rest.
  Interventions: Drug: Gemcitabine TS-1

INTERVENTIONS:
Drug: Gemcitabine TS-1 — Gemcitabine (1,000mg/m2) will be administered on days 1 and 8 at every 3 weeks TS-1 will be administered orally according to body surface area (BSA) as follows : BSA<1.25 M2, 80 mg/day; 1.25 M2≤BSA<1.5 M2, 100 mg/day; 1.5 M2≤BSA, 120 mg/day for 14 consecutive days followed by a 7-day rest.
  Other Names: Gemcitabine (Gemza)TS-1 (TS-1)

SUMMARY:
In current study, we evaluate the efficacy of gemcitabine and TS-1 combination chemotherapy in advanced BTC.

DETAILED DESCRIPTION:
At present, surgery is the only curative treatment option for biliary tract cancer (BTC). However, less than 25% of patients are resectable at presentation with high relapse rates after surgery. Because of the low incidence and heterogeneity of BTC, clinical trials are difficult to conduct in these patients, hampering the evaluation of optimal chemotherapy regimens. Owing to the lack of randomized phase III studies, there is no standard regimen for palliative chemotherapy of GBC and CC. But the exploration of an optimal regimen for standard first-line chemotherapy for BTC is imperative in order to improve survival in these patients.

Gemcitabine has demonstrated antitumor activity as monotherapy in phase II trials in BTC patients with response rates ranging from 22 to 36% (2001 Proc Am Soc Clin Oncol 20:A626, 2001 J Clin Oncol 19(20):4089-4091, 2001 Ann Oncol 12(2):183-186).

As with most gastrointestinal tumors, 5-fluorouracil (5-FU) is the most studied drug as a single agent or a combination in different dosages and schedules with response rates of 10-20% and with median survival of 7-9 months in BTC (2005 Cancer 103:111-118, 2001 Clin Cancer Res 7:3375-3380).

The combination of gemcitabine and fluoropyrimidine in biliary cancers is worthy of further evaluation. The toxicity profiles of these agents are known to be non-overlapping, and combinations have been well tolerated. Oral fluoropyrimidines are considered to be an alternative to conventional protracted 5-FU infusion as far as they provide comparable efficacy and compliance.

S-1 is oral fluoropyrimidine preparation developed by Taiho Pharmaceutical Co., Ltd. (Tokyo, Japan) that combines tegafur with two 5-FU modulators, 5-chloro-2, 4-dihydroxypyridine (CDHP) and potassium oxonate (Oxo), in a molar ratio of 1:0.4:1. Tegafur, a prodrug of 5-FU, is converted to 5-FU mainly in liver and tumor cells. CDHP, a reversible inhibitor of dihydropyrimidine dehydrogenase, suppresses the degradation of 5-FU, thereby maintaining high concentrations of 5-FU in plasma and tumor cells. CDHP also decreases cardiotoxic and neurotoxic effects by reducing the production of F-b-alanine (FBAL), the main catabolite of 5-FU. Several phase II trials showed that TS-1 monotherapy or combination with CDDP, paclitaxel or irinotecan was effective palliative treatment option for advanced gastric cancer and colorectal cancer.

In current study, we evaluate the efficacy of gemcitabine and TS-1 combination chemotherapy in advanced BTC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathologically proven, measurable, unresectable, locally advanced or metastatic adenocarcinoma arising from the intra- and extrahepatic biliary ducts or gallbladder or papilla of Vater 2. No prior chemotherapy for advanced disease was allowed 3. No concurrent radiotherapy 4. At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) 5. At least 18 years old 6. ECOG performance status of ≤ 2 7. Adequate organ function as evidenced by the following; Absolute neutophil count > 1.5 x 109/L; platelets > 100 x 109/L; hemoglobin > 10g/dL; INR ≤ 1.4; total bilirubin ≤1.5 UNL; AST and/or ALT < 5 UNL; albumin > 3g/dL or > 30µmol/L; creatinine clearance ≥ 50mL/minInformed consent signed 8. Subject able to comply with the scheduled follow-up and the management of toxicities

Exclusion Criteria:

* 1. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of TS-1 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) 2. Subject with reproductive potential (male or female) not using adequate contraceptive measures 3. Pregnancy and breast-feeding 4. Other serious illness or medical condition, notably heart or lung failure, active uncontrolled infection (infection requiring antibiotics) 5. History of significant cardiac disease, arrhythmias and angina pectoris 6. Past or concurrent history of other neoplasm, except curatively treated basal cell skin cancer or adequately treated in-situ carcinoma of the cervix 7. Other concomitant anticancer agent 8. Subjects who cannot be regularly followed up for psychological, social, familial or geographic reasons 9. Patients who are using other investigational agents or who had received investigational drugs ≤ 4 weeks prior to first study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Response rate | 1year 6months

CONTACTS AND LOCATIONS:
Overall Officials: Yeong Lim Lim, Professor, Principal Investigator — Samsung Medical Center